CLINICAL TRIAL: NCT04482231
Title: Antibiotic Observatory for Respiratory Diseases, Apart From Tuberculosis and Reportable Diseases
Acronym: AORD
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, professor semir nouira, University of Monastir
Other Study IDs: BAROMETRE
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Antibiotic Sore Tongue
Keywords: antiobiotic,; respiratory tract infections; appropriateness
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the study aimed to determine the distribution of respiratory infections in Tunisian population and evaluate the frequency of antibiotics prescribed according to current international recommendations.

DETAILED DESCRIPTION:
It is an observational, cross-sectional, multicenter, national clinical study . The study was carried out from January 2018 to August 2018 in Tunisian population involving 57 primary care outpatient centers and 6 emergency departments from the 24 departments of the country .

We included all patients with lower and upper respiratory tract infections (RTIs) who have recieved antibiotic treatment.

Lower respiratory tract infection (LRTI) include pneumonia and acute bronchitis.

Acute upper respiratory tract infection (URTIs) include rhinitis, pharyngitis/tonsillitis, and laryngitis. Rhinitis, also known as coryza, is irritation and inflammation of the mucous membrane inside the nose.

The protocol of our study includes the demographic characteristics and the history of the sample as well as the symptomatology at inclusion. The data from the clinical examination were reported by the investigating doctor. After the diagnosis retained by the doctor is noted with the management of the patient which includes additional explorations if they have been requested. Finally, the investigating doctor specifies the antibiotic therapy prescribed.Appropriateness of antibiotic prescription was assessed in patients managed in the EDs . We used the MAI score (medication appropriateness index) wich includes 10 criteria. For each criterion, the evaluator rates whether the medication is appropriate, marginally appropriate, or inappropriate. Support is provided through explicit definitions and instructions.The MAI has been used in observational and interventional studies.Its feasibility, content validity, predictive validity, and reliability have been demonstrated in ambulatory settings. The maximum score is 20 which translates into maximum inappropriateness. If a patient is on multiple drugs, this test can be repeated for each drug in order to determine a total MAI score.

ELIGIBILITY:
Inclusion Criteria:

* patients with lower and upper RTIs who recieved antibiotic treatment.

Exclusion Criteria:

* not obtained informed consent, specific respiratory infection such as tuberculosis, life-threatening emergency necessitating hospitalization or non-probabilistic antibiotic therapy and contraindication to antibiotic use

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The protocol includes the demographics, history, and the symptomatology at inclusion. After the diagnosis retained by the doctor is noted and specifies the antibiotic therapy prescribed.Appropriateness of antibiotic prescription was assessed in patients managed in the EDs. We used the MAI score (medication appropriateness index) wich includes 10 criteria. For each criterion, the evaluator rates whether the medication is appropriate, marginally appropriate, or inappropriate.If a patient is on multiple drugs, this test can be repeated for each drug.
Sampling Method: Non-Probability Sample
Enrollment: 9944 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Appropriateness of antibiotic prescription | 1 day
  dichotomous (yes / no) criterion that characterizes appropriate or inappropriate use of antibiotics based on respiratory indication and patient profile

SECONDARY OUTCOMES:
inappropriatness of antibiotic prescription | 1 day
  number of inappropriate antibiotic prescriptions by clinical indication
international recommendations | 1 day
  description of therapeutic strategies inconsistent with international recommendations
patients profile with inappropriate antibiotic therapy | 1 day
  profile of patients with inappropriate antibiotic therapy
patients profile with infectious disease | 1 day
  profile of patients with infectious disease

CONTACTS AND LOCATIONS:
Overall Officials: nouira semir, MD, Principal Investigator — University of Monastir
Locations (1):
- Emergency department of fattouma bourguiba university hospital, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bel Haj Ali K, Sekma A, Messous S, Trabelsi I, Ben Youssef J, Maghraoui H, Razgallah R, Walha A, Grissa MH, Beltaief K, Mezgar Z, Coubantini A, Bouida W, Msolli MA, Boukef R, Boubaker H, Nouira S. Appropriateness of antibiotic treatment of acute respiratory tract infections in Tunisian primary care and emergency departments: a multicenter cross-sectional study. BMC Prim Care. 2022 Nov 22;23(1):295. doi: 10.1186/s12875-022-01904-7. PMID 36418965